CLINICAL TRIAL: NCT00520767
Title: A Multicenter Phase II Trial of Bortezomib (Velcade), Melphalan, and Dexamethasone (V-MD) in Patients With Symptomatic AL-Amyloidosis or Light Chain Deposition Disease
Brief Title: Bortezomib, Melphalan, and Dexamethasone in Treating Patients With Primary Amyloidosis or Light Chain Deposition Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jeffrey Zonder, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-132; P30CA022453 (NIH); MILLENNIUM-WSU-2006-132 (Barbara Ann Karmanos Cancer Institute); WSU-HIC-060907M1F (Other: Wayne State University - Human Investigation Committee)
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Results first posted 2015-03-30 (Estimated); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Primary Systemic Amyloidosis; Light Chain Deposition Disease
Keywords: primary systemic amyloidosis; light chain deposition disease
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — Bortezomib; Dexamethasone; Calcium Dobesilate; dexamethasone 21-phosphate; dexamethasone acetate; Melphalan; Microarray Analysis; Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Melphalan, Dexamethasone, Bortezomib, (Experimental): Bortezomib 1.3 mg/m2 days 1, 8, 15, 22; Dexamethasone 40 mg/d days 1, 2, 8, 9, 15, 16, 22, 23; Melphalan 9 mg/m2/day days 1-4
  Interventions: Drug: bortezomib; Drug: dexamethasone; Drug: melphalan; Genetic: microarray analysis; Other: flow cytometry; Other: laboratory biomarker analysis; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: bortezomib — Bortezomib 1.3 mg/m2 days 1, 8, 15, 22
  Other Names: Velcade
Drug: dexamethasone — Dexamethasone 40 mg/d days 1, 2, 8, 9, 15, 16, 22, 23
  Other Names: Dexasone; Decadron; Diodex; Hexadrol; Maxidex; Dexamethasone Sodium Phosphate; Dexamethasone Acetate
Drug: melphalan — Melphalan 9 mg/m2/day days 1-4
  Other Names: Alkeran®; L-PAM; L-Sarcolysin; Phenylalanine Mustard
Genetic: microarray analysis — ≤28 days prior to enrollment
Other: flow cytometry — Day 1 of cycles 6, 12, 18 and at end of study.
Other: laboratory biomarker analysis — ≤28 days prior to enrollment
Procedure: quality-of-life assessment — Start of each cycle

SUMMARY:
RATIONALE: Giving bortezomib together with melphalan and dexamethasone may be an effective treatment for primary amyloidosis and light chain deposition disease.

PURPOSE: This phase II trial is studying how well giving bortezomib together with melphalan and dexamethasone works in treating patients with primary amyloidosis or light chain deposition disease.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the complete hematologic response rate at 12 months.

Secondary

* Determine the overall hematologic response rate.
* Determine the organ response rate.
* Determine time to treatment failure.
* Determine the overall survival.

OUTLINE: This is a multicenter study.

Patients receive oral melphalan on days 1-4, bortezomib IV on days 1, 8, 15, and 22, and dexamethasone orally or IV on days 1, 2, 8, 9, 15, 16, 22, and 23. Treatment repeats every 4-6 weeks for up to 20 courses in the absence of disease progression or unacceptable toxicity.

Blood, urine, and bone marrow aspirates are collected at baseline and periodically after treatment to permit the correlation of clinical results with measured molecular events. A single baseline peripheral blood DNA sample is collected for future association studies linking disease onset, progression, and response to administered therapy with single nucleotide polymorphisms. Blood plasma and urine samples are evaluated for proteomic markers associated with disease progression and therapeutic response. Peripheral blood RNA samples are evaluated for transcriptional response to treatment of peripheral blood lymphocytes. Bone marrow aspirates are collected to extract plasma cells by flow cytometry for gene expression profiling.

Quality of life is assessed at the beginning of each course.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy-proven diagnosis of 1 of the following:

  * Primary systemic amyloidosis

    * Histochemical diagnosis of amyloidosis determined by polarizing microscopy of green bi-refringent material in Congo red-stained tissue specimens or characteristic electron microscopy appearance
  * Light chain deposition disease
* Measurable disease as defined by one or more of the following:

  * Serum monoclonal protein ≥ 0.5 g/dL by serum electrophoresis
  * Urine monoclonal protein > 200 mg/tv in a 24 hr urine electrophoresis
  * Serum immunoglobulin free-light chain ≥ 10 mg/dL AND abnormal serum immunoglobulin kappa lambda free light chain ratio
* Must meet 1 of the following criteria:

  * Clonal population of plasma cells in the bone marrow (≤ 30%)
  * Immunohistochemical stain with anti-light chain anti-sera of amyloid fibrils
* Must not meet the following diagnostic criteria for symptomatic* multiple myeloma:

  * Lytic lesions on skeletal survey
  * Plasmacytoma
  * Increase in bone marrow plasma cells ≥ 30% NOTE: *Patients who meet the International Myeloma Working Group definition of symptomatic multiple myeloma with symptoms attributable only to associated amyloidosis and who do not otherwise meet the criteria for diagnosis of smoldering myeloma are potentially eligible upon approval of the principal investigator.
* If not previously treated, patient is either not a candidate for autologous stem cell transplantation (ASCT) or has declined the option of ASCT

  * Patients who have undergone prior ASCT and have subsequently progressed are eligible, provided other eligibility criteria are met
* No secondary or familial amyloidosis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-3
* Creatinine < 5 mg/dL
* Bilirubin < 2.5 times upper limit of normal (ULN)
* ALT and AST < 3 times ULN
* Absolute neutrophil count ≥ 1,000/mm³
* Platelet count ≥ 80,000/mm³
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Peripheral sensory neuropathy < grade 3
* No myocardial infarction within the past 6 months
* No New York Heart Association class III or IV heart failure
* No uncontrolled angina
* No severe uncontrolled ventricular arrhythmias
* No EKG* evidence of acute ischemia or active conduction system abnormalities (not including 1st degree AV-block, Wenckebach type 2nd degree heart block, or left bundle branch block) NOTE: *Prior to study entry, any EKG screening abnormality must be documented by the investigator as not medically relevant; there is no lower limit of LVEF below which patients are excluded from participation
* No hypersensitivity to bortezomib, boron, or any of the other agents utilized in this study
* No serious concurrent illness (e.g., stroke) within the past 30 days
* No psychiatric illness likely to interfere with study participation
* No untreated HIV infection

  * Patients with asymptomatic HIV infection on active antiretroviral therapy are potentially eligible
* No diagnosis or treatment of another malignancy within the past 3 years, except completely resected basal cell or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No other investigational drugs within the past 14 days

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-09; Primary Completion 2010-10 (Actual); Study Completion 2019-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Zonder, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (7):
- United States (7):
  - Rocky Mountain Cancer Centers/Rocky Mountain Blood & Marrow Transplant Program, Denver, Colorado
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Melphalan, Dexamethasone, Bortezomib,
Started | 35
Completed | 33
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Melphalan, Dexamethasone, Bortezomib,
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 64 [47 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Complete Hematologic Response
Time Frame: Up to 12 months
Population: Individuals evaluable for response
Measure: Number; unit: participants
Arm/Group | Melphalan, Dexamethasone, Bortezomib,
Number analyzed (Participants) | 33
participants | 16

2. Secondary Outcome: Overall Survival
Description: time from day of registration until day of death.
Time Frame: time from day of registration until 72 months.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Melphalan, Dexamethasone, Bortezomib,
Number analyzed (Participants) | 35
month | 31.1 [22.1 to 45.5]

3. Secondary Outcome: Time to Treatment Failure (TTF)
Description: Time from start of treatment until date of documented disease progression, removal from protocol due to toxicity, or death from any cause.
Time Frame: start of treatment until 72 months
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Melphalan, Dexamethasone, Bortezomib,
Number analyzed (Participants) | 35
month | 18.1 [10.8 to 34.4]

4. Secondary Outcome: Organ Response Rate (OrR)
Time Frame: Beginning of cycles 4, 8, 12, 16 and 20, at follow up and end of study.
Population: Not collected not analyzed.
Arm/Group | Melphalan, Dexamethasone, Bortezomib,
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Hematologic Response Rate (OHR)
Time Frame: Beginning of cycles 4, 8, 12, 16 and 20, at follow up and end of study.
Population: Not collected not analyzed.
Arm/Group | Melphalan, Dexamethasone, Bortezomib,
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Melphalan, Dexamethasone, Bortezomib,
Serious Adverse Events (participants affected / at risk) | 12/35
Other Adverse Events (participants affected / at risk) | 3/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melphalan, Dexamethasone, Bortezomib, (N=35)
Death (General disorders) | 2 (2)
Infection with Normal ANC-Lung (pneumonia) (Infections and infestations) | 2 (2)
Pain-chest wall (General disorders) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Mental Status Change (Psychiatric disorders) | 2 (2)
Hypotension (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Creatinine (Metabolism and nutrition disorders) | 2 (2)
Ventricular Arrhythmia (Cardiac disorders) | 2 (2)
Edema (Blood and lymphatic system disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
syncope (Nervous system disorders) | 1 (1)
Hypertension (Cardiac disorders) | 2 (2)
Pain-Headache (Nervous system disorders) | 2 (2)
Renal Failure (Renal and urinary disorders) | 1 (1)
Infection with Normal ANC-Catheter related (Infections and infestations) | 1 (1)
Infection with Normal ANC-Skin (cellulitis)-shingles (Infections and infestations) | 1 (1)
cardiac Arrhythmia (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melphalan, Dexamethasone, Bortezomib, (N=35)
Constipation (Gastrointestinal disorders) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Mix of previously treated & newly diagnosed pts (populations which may have different prognoses), plus the relatively small trial size limit conclusions one can draw re: relative efficacy of MDV (vs CyBorD or Mel-Dex, for example)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No